CLINICAL TRIAL: NCT06521177
Title: A Trial to Examine the Efficacy of a Hand Serum and Glove Combination.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Habelo Beauty (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20418
Record Dates: First submitted 2024-07-17; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Skin Health; Dermatology; Skin Care
Keywords: Cosmetic Study; Anti-Aging; Skin Appearance
MeSH Terms: interventions — Gloves, Protective

STUDY DESIGN:
Intervention Model Description: A crossover trial where participants are randomized to receive either Hand Serum alone or Hand Serum with Glove in the first period, followed by the alternate intervention in the second period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand Serum Alone First (Experimental): Participants will apply Hand Serum alone for the first period (6 weeks), followed by applying Hand Serum with Glove in the second period (6 weeks).
  Interventions: Other: Hand Serum and Glove
- Hand Serum with Glove First (Experimental): Participants will apply Hand Serum with Glove for the first period (6 weeks), followed by applying Hand Serum alone in the second period (6 weeks).
  Interventions: Other: Hand Serum and Glove

INTERVENTIONS:
Other: Hand Serum and Glove — Participants will apply the Hand Serum to both hands daily for 8 weeks. During Weeks 7-8, participants will also wear a glove on one hand. The intervention aims to improve skin health and appearance on the hands, assessed through questionnaires and expert skin grading.

SUMMARY:
This is a virtual, 8-week, interventional crossover trial with 33 female participants aged 35 and older. The study aims to evaluate the efficacy of Habelo Beauty's Activating Hand Serum and Glove combination in improving hand skin health and appearance. During Weeks 1-6, participants will apply the Hand Serum to both hands daily. In Weeks 7-8, they will continue applying the Hand Serum and also wear a glove on one hand. Assessments will be conducted via questionnaires and photos at multiple time points to evaluate primary and secondary endpoints related to skin health parameters.

ELIGIBILITY:
Inclusion Criteria:

* Female, 35+ years old.
* Concerns about signs of skin aging on hands.
* Willing to discontinue other hand lotions or serums.
* Generally healthy, able to follow the study protocol.
* Access to someone to take hand photos at Baseline and Week 8.
* Consistent use of SPF for the duration of the study.

Exclusion Criteria:

* Chronic skin conditions on hands.
* History of skin cancer or pre-cancerous lesions on hands.
* Pregnant, breastfeeding, or trying to conceive.
* Inability to follow study protocol.
* Current significant medical procedures planned within the study duration.
* Severe allergies or reactions to product ingredients.
* Current or planned hand casting or splinting.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
Improvement in Overall Skin Health and Hydration using Expert Skin Grading | Baseline, Day 1, Week 2, Week 4, Week 6, and Week 8
  Assessment of overall skin health and hydration parameters, measured through expert skin grading and study-specific questionnaires. These assessments will be conducted at Baseline, Day 1, Week 2, Week 4, Week 6, and Week 8.
Improvement in Skin Radiance and Plumpness using Expert Skin Grading | Baseline, Day 1, Week 2, Week 4, Week 6, and Week 8
  Assessment of skin radiance and plumpness parameters, measured through expert skin grading and study-specific questionnaires. These assessments will be conducted at Baseline, Day 1, Week 2, Week 4, Week 6, and Week 8.
Reduction in Dark Spots and Redness using Expert Skin Grading | Baseline, Day 1, Week 2, Week 4, Week 6, and Week 8
  Assessment of dark spots and redness, measured through expert skin grading and study-specific questionnaires. These assessments will be conducted at Baseline, Day 1, Week 2, Week 4, Week 6, and Week 8.
Reduction in Fine Lines and Crepe Appearance using Expert Skin Grading | Baseline, Day 1, Week 2, Week 4, Week 6, and Week 8
  Assessment of fine lines and 'crepe' appearance, measured through expert skin grading and study-specific questionnaires. These assessments will be conducted at Baseline, Day 1, Week 2, Week 4, Week 6, and Week 8.

SECONDARY OUTCOMES:
Participant Perception of Skin Health and Appearance Between Gloved and Non-Gloved Hand using Study-Specific Perception Questionnaire | Baseline and Week 8
  Comparison of participant perception of skin health and appearance changes between the hand that had the Hand Serum only applied and the hand that had the Hand Serum plus the Glove at Endline. This will be assessed via a study-specific perception questionnaire at Baseline and Endline.
Expert Skin Grading of Skin Health and Appearance Between Gloved and Non-Gloved Hand | Baseline and Week 8
  Comparison of expert skin grading of skin health and appearance changes between the hand that had the Hand Serum only applied and the hand that had the Hand Serum plus the Glove at Endline. This will be conducted at Baseline and Endline.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No